CLINICAL TRIAL: NCT03527927
Title: sTep dOWn Inhalers in the reAl woRlD
Acronym: TOWARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hywel Dda Health Board (Other)
Collaborators: Swansea University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HywelDdaHB
Record Dates: First submitted 2018-04-18; First posted 2018-05-17 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LABA/LAMA inhaler (Experimental): Patients on a combination of inhaled corticosteroid (ICS), long acting beta agonist (LABA) and long acting muscarinic antagonist (LAMA) will be taken off their current ICS/LABA/LAMA combination inhalers and will commence on a single LABA/LAMA inhaler (any LABA/LAMA) of their choice.
  Interventions: Drug: Any LABA/LAMA

INTERVENTIONS:
Drug: Any LABA/LAMA — Following consent, patients will be taken off their current ICS/LABA/LAMA combination inhalers and shown 4 single inhaler LABA/LAMA devices and asked to choose a preferred device to use, provided they can demonstrate effective use.
  Other Names: Long acting beta agonist; Long acting muscarinic antagonist

SUMMARY:
To establish the feasibility of stopping inhaled steroids and switching or maintaining dual bronchodilation in one visit - in the real world, for people with COPD.

DETAILED DESCRIPTION:
COPD patients prescribed a combination of any inhaled corticosteroid (ICS), long acting beta agonist (LABA) and long acting muscarinic antagonist (LAMA) will be switched to a single LABA/LAMA combination inhaler, stopping their ICS. They will be followed up for 12 months.

Participants are shown the four currently available LABA/LAMA combination inhalers and instructed on their use. The clinical specialist will use standard prompts in an effort to demonstrate the inhalers in an unbiased way. The participants will choose: Ultibro® (Breezhaler device) or Duaklir® (Genuair device) or Anoro® (Ellipta device) or Spiolto® (Respimat device) and they will be prescribed the inhaler of their choice provided they can demonstrate effective use.

Patients will be reviewed 4, 12, 26 and at 52 weeks after switching with clinical outcomes measured at these points. As this is a real-world open study the patients and GPs are instructed that treatments can be changed at any point as clinically indicated, including restarting an ICS.

ELIGIBILITY:
Inclusion Criteria:

* GP diagnosis of COPD
* Post bronchodilator FEV1/FVC ratio <70% with FEV1<80% predicted
* Current or ex smoker equal or greater than 10 pack years
* Taking an ICS, LABA & LAMA

Exclusion Criteria:

* Unable or unwilling to sign informed consent
* Any previous or current diagnosis of asthma
* Any features of asthma or large variability in symptoms
* History of atopy
* Any previous blood eosinophil count >600mm3
* A moderate or severe exacerbation of COPD (needing systemic glucocorticosteroids or hospital admission for >24 hours) within the last 6 weeks
* Life expectancy < 1 year

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Numbers maintained on dual bronchodilation | At 12 months
  The proportion of patients with stable COPD who can be successfully switched from triple inhaled therapy (ICS+LABA+LAMA in any combination of inhalers) to dual inhaled bronchodilator therapy (LABA+LAMA)

SECONDARY OUTCOMES:
Moderate or severe exacerbations | 12 months before and 12 months after enrollment
  Comparison of the number of moderate and severe exacerbations in those on LABA+LAMA over 52 weeks compared with their previous 52 weeks
Exacerbations | 12 months before and 12 months after enrollment
  Comparison of the number of moderate and severe exacerbations in those on LABA+LAMA over 52 weeks compared with those continuing triple therapy
Restarting inhaled steroids | At 12 months
  Proportion of patients requiring restarting ICS (on the discretion of their clinician) at each visit.
Lung function | Baseline, 4 weeks, 12 weeks, 26 weeks, 52 weeks
  Trend in FEV1
COPD assessment test (CAT) | Over 12 months
  Changes in total CAT score (range 0-40), higher score indicates worse outcome) from baseline, at 4 weeks, 12 weeks, 26 weeks and 52 weeks
Costs | 12 months before and 12 months after enrollment
  Comparison of total inhaler prescription costs
Inhaler device choice | At enrollment
  Proportions of patients choosing each LABA+LAMA device and some reasons why
EQ-5D-3L | Over 12 months
  General quality of life visual analogue scale from 0-100, 0 indicates worse imaginable health and 100 best imaginable health. Score reported at baseline, 4 weeks, 12 weeks, 26 weeks and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Keir E Lewis, Prof, Study Director — Hywel Dda University Health Board
Locations (1):
- Prince Philip Hospital, Llanelli, Carmarthenshire, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT03527927/Prot_000.pdf